CLINICAL TRIAL: NCT06895174
Title: Efficacy Of Mandibular Parasymphysis Fracture Treatment With Two Miniplates Versus One Miniplate With Arch Bar
Brief Title: Comparison of the Post-operative Efficacy of Arch Bar With Single Plate and Two Plate Fixation in Mandibular Parasymphsis Fracture.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: HITEC-Institute of Medical Sciences (Other)
Responsible Party: Principal Investigator, Fatima Khattak, Assistant Professor Oral & Maxillofacial Surgery, HITEC-Institute of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: fatimakhattak12@gmail.com
Record Dates: First submitted 2025-03-24; First posted 2025-03-26 (Actual); Last update posted 2025-10-08 (Actual); Status verified 2024-07

CONDITIONS: Mandible Fracture
MeSH Terms: conditions — Mandibular Fractures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Titanium miniplates (Active Comparator): Titanium miniplates are used in open reduction and internal fixation for facial fractures including mandible fractures.One miniplate is placed on superior border and other is placed at inferior border for mandible parasymphysis fracture.
  Interventions: Device: Titanium miniplates
- Arch bars (Other): One Arch bar placed in tension zone for closed reduction technique in mandible fractures is combined with single miniplate placed at the lower border and its efficacy will be compared with two miniplates group
  Interventions: Other: Arch Bar

INTERVENTIONS:
Device: Titanium miniplates — Titanium miniplates are used for open reduction and internal fixation in mandible fractures according to Champy's principle of osteosynthesis
  Arms: Titanium miniplates
Other: Arch Bar — Arch bars are used for intermaxillary fixation in facial fractures as a mean of closed reduction.In this study arch bars placed in tension zone will be combined with single miniplate placed at inferior border of mandible and this modality efficacy will be compared with two miniplate group.
  Arms: Arch bars

SUMMARY:
This clinical trial is designed to compare post-operative infection, symptoms of paresthesia, inferior border misalignment and operating time of one plate with arch bar against standard two miniplates in mandibular parasymphysis fracture in order to achieve the treatment which is beneficial for the patients. This study will contribute to literature for the betterment of patient.

The objective of this study is to compare the post-operative efficacy of arch bar with single plate and two plate fixation in mandibular parasymphsis fracture.

ELIGIBILITY:
Inclusion Criteria:

* All patients with mandibular unilateral parasymphysis fracture

Exclusion Criteria:

1. Mandibular defect fractures.
2. Grossly comminuted fractures.
3. Medically compromised patient.(e.g uncontrolled metabolic disease

   * immunocompromised patient, patient receiving radiation and chemotherapy).
4. Multiple fracture of Mandible.

Ages: 17 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Osseous alignment | Final Alignment will be checked after one month
  It is checked after the surgical procedure by evaluating the continuity of lower border of mandible on orthopentomogram on first post-operative day, after 15 days and after 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Dental College Hitec Institute Of Medical Sciences Taxila Cantt, Taxila, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided
it is not required for this study